CLINICAL TRIAL: NCT01503346
Title: Taking Herbal Formula：DaHuang GangTsao Tang to Improve the Appetite Loss Condition of Cancer Patients in Late-stage：A Clinical Control Trial Study
Brief Title: DaHuang GangTsao Tang to Improve the Appetite Loss Condition of Cancer Patients
Acronym: TCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 100610; Protocol Record 100610 (Registry Identifier: YDLiu)
Record Dates: First submitted 2011-11-07; First posted 2012-01-04 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Non-organic Loss of Appetite
Keywords: Appetite Loss
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- herbal medicine (Experimental): Intervention group
  * 1. 2 grams of DaHuang abstract powder and 0.5 grams GanTsao abstract powder are mixed and separated into four packages;
  * 2. each package was given to each patient four times a day (three time after meal and one time before sleep);
  * 3. each patient received the usual medication of the hospice ward at the same time;
  * 4. record the patients' score of pre-test, mid-test and after-test of QIPCTP at the 1st day, the 3rd day and the 6th day;
  * 5. record the patients' score of EORTC QLQ-C30 V3.0 and ECOG (Eastern Cooperative Oncology Group Performance Status) at the 1st day and the 6th day.
  Interventions: Drug: DaHuang GanTsao Tang

INTERVENTIONS:
Drug: DaHuang GanTsao Tang — Intervention group
  1. 2 grams of DaHuang abstract powder and 0.5 grams GanTsao abstract powder are mixed and separated into four packages;
  2. each package was given to each patient four times a day (three time after meal and one time before sleep);
  3. each patient received the usual medication of the hospice ward at the same time;
  4. record the patients' score of pre-test, mid-test and after-test of QIPCTP at the 1st day, the 3rd day and the 6th day;
  5. record the patients' score of EORTC QLQ-C30 V3.0 and ECOG (Eastern Cooperative Oncology Group Performance Status) at the 1st day and the 6th day.
  Other Names: Herbal Medicine Group

SUMMARY:
Appetite loss is a severe and common symptom among late-stage cancer patients, and it causes great the anxiety for the patient's family. In TCM theory, the investigators call these patients are in block and repulsion condition. The investigators try to set a study to use the herbal medicine solution taken in frequent small amounts by cancer patients in late-stage to improve the appetite loss condition. Through this method, the investigators not only want to improve the quality of life of cancer patients in late-stage but also set a valuable treatment.

DETAILED DESCRIPTION:
Intervention group

* 1. 2 grams of DaHuang abstract powder and 0.5 grams GanTsao abstract powder are mixed and separated into four packages;
* 2. each package was given to each patient four times a day (three time after meal and one time before sleep);
* 3. each patient received the usual medication of the hospice ward at the same time;
* 4. record the patients' score of pre-test, mid-test and after-test of QIPCTP at the 1st day, the 3rd day and the 6th day;
* 5. record the patients' score of EORTC QLQ-C30 V3.0 and ECOG (Eastern Cooperative Oncology Group Performance Status) at the 1st day and the 6th day.

Control group

* 1. each patient received the usual medication of the hospice ward during the trial interval;
* 2. record the patients' score of receive pre-test, mid-test and after-test of QIPCTP at the 1st day, the 3rd day and the 6th day;
* 3. record the patients' score of EORTC QLQ-C30 V3.0 and ECOG (Eastern Cooperative Oncology Group Performance Status) at at the 1st day and the 6th day.

Medicine DaHuang herbal abstract powder is produced by Sun Ten Pharmaceutical Co., Ltd, and it's product serial number: 276001. GanCao herbal abstract powder is also produced by Sun Ten Pharmaceutical Co., Ltd, and it's product serial number: 185645. Each herbal abstract powder is qualified with the data of HPLC to confirm each content and stability. The pharmaceutical company is qualified by Good Manufacturing Practice (GMP) certification in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Terminal cancer patients in hospice ward
* Patients with appetite loss condition
* Ages between 20 to 80 years old
* No history of diabetes

Exclusion Criteria:

* Entered the stage of dying patients
* Receiving other traditional Chinese medicine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
appetite score | 6 days
  The investigators detect the patients' appetite condition at the 1st,3rd and 6th day.

CONTACTS AND LOCATIONS:
Overall Officials: Yu De LIU, Master, Study Chair — Changhua Christian Hospital
Locations (1):
- Changhua Christan Hospital, Changhua, Changhua Country, Taiwan